CLINICAL TRIAL: NCT04009837
Title: Manual Therapy and Strengthening for the Hip in Older Adults With Chronic Low Back Pain (MASH): A Randomized Clinical Trial
Brief Title: Manual Therapy and Strengthening for the Hip in Older Adults With Chronic Low Back Pain
Acronym: MASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: University of Pittsburgh (Other); Duke University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Gregory Evan Hicks, Professor, Chair of the Department of Physical Therapy, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1210486; R01AG041202-06 (NIH)
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Results first posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Chronic Low-back Pain; Hip Impairments; Hip-spine Syndrome; Osteoarthritis
Keywords: older adult; geriatrics; chronic low back pain; low back pain; hip-spine; rehabilitation; physical therapy; spine; hip pain
MeSH Terms: conditions — Osteoarthritis; Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip-focused (Experimental): Hip-focused rehabilitation intervention
  Interventions: Behavioral: Hip-focused rehabilitation intervention
- Spine-focused (Active Comparator): Spine-focused rehabilitation intervention
  Interventions: Behavioral: Spine-focused rehabilitation intervention

INTERVENTIONS:
Behavioral: Hip-focused rehabilitation intervention — The hip-focused intervention includes a blend of hip-focused rehabilitative techniques and some basic lumbar spine-directed techniques. The hip-focused arm includes tailored manual therapy, progressive strengthening exercises, and flexibility exercises for the hip, as well as spinal flexibility and trunk muscle training exercises. The intervention will be delivered by licensed physical therapists in one-hour sessions, twice per week, for 8 weeks.
  Arms: Hip-focused
Behavioral: Spine-focused rehabilitation intervention — The spine-focused rehabilitation intervention is a direct and comprehensive lumbar spine rehabilitative program, but it does not include hip treatment. The spine-focused arm includes spinal manual therapy, spinal flexibility exercises, and trunk muscle training exercises. The intervention will be delivered by licensed physical therapists in one-hour sessions, twice per week, for 8 weeks.
  Arms: Spine-focused

SUMMARY:
Older adults with chronic low back pain (LBP) are at a greater risk for disability, loss of independence, and lower quality of life. Experts agree that LBP is not a homogeneous condition, and treatments should differ based upon clinical presentation. Our past work indicates that all of these hip and lumbar spine impairments may contribute to worse physical function and greater disability, but the relative importance of each impairment is unclear. Thus, clinicians have limited evidence to draw on for treatment decisions for this patient population. We have identified a vulnerable subgroup of older adults with hip and low back pain. The purpose of this study is to randomize participants into one of two treatment arms and analyze the outcomes.

DETAILED DESCRIPTION:
This randomized clinical trial is designed to explore two different interventions: one that addresses these hip issues (hip-focused) and one that focuses more directly on the lumbar spine (spine-focused). We aim to recruit a sample of 180 older adults who have chronic LBP and hip impairments (i.e. pain and muscle weakness). To ensure our findings are generalizable, the study will be conducted across three sites in different geographical regions: University of Delaware, University of Pittsburgh, and Duke University.

The goal of this clinical trial is to learn more about how older adults with low back and hip pain respond to physical therapy intervention.

Participants will have three standardized assessments by licensed physical therapists, at baseline, 8 weeks, and 6 months. Once randomized, participants will attend on-site sessions 2x per week for 8 weeks and complete a home exercise log. People in the hip-focused group will receive mobilizations and stretching, and will participate in hip exercises and trunk muscle exercise. People in the spine-focused group will receive massage and gentle mobilizations to the lumbar spine and participate in stationary cycling and trunk muscle training.

ELIGIBILITY:
Inclusion Criteria:

* LBP duration ≥ 3 months
* LBP an ongoing problem for at least half days in past 6 months
* LBP intensity > 3 on scale of 0 (no pain) to 10 (worst pain imaginable)
* Classified into the "weak+painful" hip-spine subgroup based on two criterion. Participants must have: 1) hip internal rotation strength (normalized to body weight) in at least one hip that is < 0.26; and, 2) from the Hip Disability and Osteoarthritis Outcome Score (HOOS) Pain items P4-P8, a raw score sum of >5 (0-20 range, where higher scores indicate more pain interference with daily activities).

Exclusion Criteria:

* Previous hip fracture with surgical repair
* Previous hip fracture without surgical repair within the past 15 years
* Total hip replacement
* Known spinal pathology other than osteoarthritis (e.g. recent back surgery, vertebral fractures in the past year, rheumatoid arthritis, metastases)
* Non-ambulatory or severely impairment mobility (i.e. requires wheelchair)
* Folstein Mini-Mental State Examination score of < 24, indicating cognitive impairment
* Severe visual or hearing impairment
* Unable to read or speak English
* Red flags indicative of serious disorder underlying LBP (e.g. fever associated with LBP, significant unintentional weight loss > 10 pounds, pain that awakes or keeps one awake at night)
* Significant pain the legs greater than the back
* Acute illness (e.g. hospitalization within the past 3 months or current infection)
* Inability to participate in study for the full six months for any known reason
* Received physical therapy for low back or hip within the last 3 months

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory E Hicks, PhD, Principal Investigator — University of Delaware
Locations (3):
- United States (3):
  - University of Delaware, Newark, Delaware
  - Duke University, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Hicks GE, George SZ, Pugliese JM, Coyle PC, Sions JM, Piva S, Simon CB, Kakyomya J, Patterson CG. Hip-focused physical therapy versus spine-focused physical therapy for older adults with chronic low back pain at risk for mobility decline (MASH): a multicentre, single-masked, randomised controlled trial. Lancet Rheumatol. 2024 Jan;6(1):e10-e20. doi: 10.1016/S2665-9913(23)00267-9. PMID 38258673
- [Derived] Pugliese JM, Coyle PC, Knox PJ, Sions JM, Patterson CG, Pohlig RT, Simon CB, Weiner DK, George SZ, Piva S, Hicks GE. The Manual Therapy and Strengthening for the Hip (MASH) Trial: Protocol for a Multisite Randomized Trial of a Subgroup of Older Adults With Chronic Back and Hip Pain. Phys Ther. 2022 Jan 1;102(1):pzab255. doi: 10.1093/ptj/pzab255. PMID 34751784

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Older adults aged 60-85 with chronic low back pain and hip pain were recruited from communities in Newark, Delaware; Pittsburgh, Pennsylvania; and Durham, North Carolina. Recruitment (from November 1, 2019 through April 30, 2022) included newspaper advertisements, visits to senior centers, clinic referrals, research registries, and electronic medical records.
Period: Overall Study
Arm/Group | Hip-focused | Spine-focused
Started | 91 | 93
8-Weeks (Post-intervention) | 83 | 82
Completed | 83 | 82
Not Completed | 8 | 11
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Did not complete any aspect of of 8-week assessment | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hip-focused | Spine-focused | Total
Number analyzed (Participants) | 91 | 93 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (6.0) | 70.6 (6.4) | 70.71 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 60 | 121
  Male | 30 | 33 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 90 | 92 | 182
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 15 | 32
  White | 72 | 77 | 149
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 91 | 93 | 184
Low Back Pain duration (years) [Mean (Standard Deviation); unit: years] | 15.7 (14.6) | 14.0 (12.0) | 14.8 (13.4)

OUTCOME MEASURES:

1. Primary Outcome: Quebec Back Pain Disability Scale
Description: A 20-item questionnaire that assesses limitations in daily activities due to back pain. Scores can range from 0-100% with higher scores indicating greater back pain-related disability.
Time Frame: Baseline to 8-week assessment (i.e. post-intervention)
Population: The number analyzed in one or more rows differs from the overall number analyzed because some participants withdrew from the study over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
score on a scale
  Baseline | 27.9 (15.8) | 27.9 (15.5)
  8-weeks (post-intervention): number analyzed (Participants) | 83 | 82
  8-weeks (post-intervention) | 16.7 (11.7) | 20.3 (14.3)

2. Primary Outcome: 10-Meter Walk Test at Self-Selected Speed (10MWT)
Description: A performance test where participants walk along a 10-meter linear pathway at their 'usual pace' for three trials. Average self-selected gait speed is determined over the central 6 meters of the course in meters/second. Faster walking speeds indicate better mobility.
Time Frame: Baseline to 8-week assessment (i.e. post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
meters/second
  Baseline | 1.12 (0.25) | 1.12 (0.24)
  8-week (post-intervention) assessment: number analyzed (Participants) | 81 | 82
  8-week (post-intervention) assessment | 1.2 (0.24) | 1.21 (0.23)

3. Secondary Outcome: Quebec Back Pain Disability Scale
Description: as for outcome 1
Time Frame: Baseline to the 6-month assessment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
score on a scale
  Baseline | 27.9 (15.8) | 27.9 (15.5)
  6-months (final assessment): number analyzed (Participants) | 83 | 79
  6-months (final assessment) | 15.8 (12.5) | 17.3 (14.1)

4. Secondary Outcome: 10 Meter Walk Test -- Self-Selected Gait Speed at 6 Months (Final Assessment)
Description: as for outcome 2
Time Frame: Baseline to 6-months
Population: The number analyzed in some rows differs from overall number analyzed as some participants withdrew from the study over time.
Measure: Mean (Standard Deviation); unit: Meters/second
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
Meters/second
  Baseline | 1.12 (0.25) | 1.12 (0.24)
  6-months: number analyzed (Participants) | 76 | 74
  6-months | 1.21 (0.25) | 1.24 (0.22)

5. Secondary Outcome: 10-Meter Walk Test at Fast Speed (10MWT)
Description: A performance test where participants walk along a 10-meter linear pathway 'as quickly as possible', for three trials. Average fast gait speed is determined over the central 6 meters of the course in meters/second. Faster walking speeds indicate better mobility.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
meters/second
  Baseline | 1.57 (0.34) | 1.59 (0.38)
  8-weeks (post-intervention): number analyzed (Participants) | 78 | 78
  8-weeks (post-intervention) | 1.65 (0.31) | 1.67 (0.32)
  6-months (final assessment): number analyzed (Participants) | 71 | 69
  6-months (final assessment) | 1.63 (0.31) | 1.66 (0.34)

6. Secondary Outcome: Timed Up-and-Go (TUG)
Description: A performance test where participants rise from a chair, walk 3 meters at their regular pace, and return to a seated position in the same chair. One practice trial is performed followed by three timed trials; performance times are averaged. Greater times indicate worse physical function.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
Seconds
  Baseline | 9.73 (2.68) | 9.46 (2.07)
  8-weeks (post-intervention): number analyzed (Participants) | 78 | 77
  8-weeks (post-intervention) | 8.92 (1.89) | 9.12 (1.93)
  6-months (final assessment): number analyzed (Participants) | 71 | 69
  6-months (final assessment) | 8.99 (1.93) | 8.82 (2.03)

7. Secondary Outcome: Six-Minute Walk Test (6MWT)
Description: A performance test where participants are asked to walk as far as they can in six minutes around a continuous track. Greater distances (in meters) indicate better mobility and exercise tolerance.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 89 | 93
Meters
  Baseline | 451.0 (116.7) | 451.9 (101.6)
  8-weeks (post-intervention): number analyzed (Participants) | 78 | 75
  8-weeks (post-intervention) | 489.0 (100.4) | 468.2 (108.8)
  6-months (final assessment): number analyzed (Participants) | 67 | 69
  6-months (final assessment) | 487.8 (100.1) | 477.9 (105.9)

8. Secondary Outcome: 30 Second Chair Stand Test
Description: A performance test where participants perform as many sit-to-stands as possible in 30 seconds while their arms are folded across their chest. The number of stands are counted. Higher numbers correlate with better scores.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of repetitions
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 89 | 93
number of repetitions
  Baseline | 10 (3.7) | 10 (3.2)
  8-weeks (post-intervention): number analyzed (Participants) | 80 | 80
  8-weeks (post-intervention) | 11 (3.1) | 11 (3.3)
  6-months (final assessment): number analyzed (Participants) | 71 | 73
  6-months (final assessment) | 12 (3.4) | 11 (3.8)

9. Secondary Outcome: Movement-evoked Pain From the 6MWT and the 30 Second Chair Stand Test
Description: Post-test pain intensities, i.e., 0-10, for both the Six-Minute Walk Test and the 30 Second Chair Stand Test were used in the calculation of aggregate movement-evoked pain. Scores for this measure were the sum of both post-test pain intensities, resulting in a score range of 0-20, where higher numbers indicate worse pain.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 89 | 93
score on a scale
  Baseline | 6.4 (4.3) | 6.7 (4.7)
  8-weeks (post-intervention): number analyzed (Participants) | 78 | 75
  8-weeks (post-intervention) | 3.6 (3.6) | 5.2 (4.5)
  6-months (final assessment): number analyzed (Participants) | 68 | 69
  6-months (final assessment) | 3.8 (4.1) | 4.1 (4.1)

10. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: A 9-item questionnaire that assesses the presence/absence of depressive symptoms. Scores above 5 indicate likeliness of depressive symptoms. Scores range from 0-27.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: The number analyzed in one or more rows differs from overall number analyzed because some participants withdrew from the study over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
score on a scale
  Baseline | 3.3 (4.1) | 2.9 (3.6)
  8 week (post-intervention): number analyzed (Participants) | 83 | 83
  8 week (post-intervention) | 2.5 (2.7) | 2.6 (3.6)
  6 months (final assessment): number analyzed (Participants) | 83 | 79
  6 months (final assessment) | 2.4 (2.8) | 2.5 (3.5)

11. Secondary Outcome: Low Back Activity Confidence Scale (LOBACS)
Description: A 15-item questionnaire that measures a person's confidence in their ability to perform different activities, including carrying, pushing, sitting, walking, and exercising, which may be directly affected by low back pain. There is an overall score, as well as three Self-Efficacy Subscales: Functional, Self-Regulatory, and Exercise. Overall, as well as subscales, range from 0-100%, where higher numbers indicate higher confidence.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
score on a scale
  Baseline: Overall | 70.1 (16.4) | 68.9 (18.8)
  8-week: Overall: number analyzed (Participants) | 83 | 83
  8-week: Overall | 78.4 (14.9) | 74.3 (19.9)
  6-month: Overall: number analyzed (Participants) | 83 | 79
  6-month: Overall | 76.2 (18.8) | 73.0 (20.3)
  Baseline: Functional Subscale | 56.2 (23.9) | 54.3 (23.4)
  8-week: Functional Subscale: number analyzed (Participants) | 83 | 83
  8-week: Functional Subscale | 68.2 (21.1) | 63.1 (26.0)
  6-month: Functional Subscale: number analyzed (Participants) | 83 | 79
  6-month: Functional Subscale | 70.0 (23.9) | 65.2 (25.6)
  Baseline: Self-Regulatory Subscale | 78.4 (19.1) | 77.9 (23.6)
  8-week: Self-Regulatory Subscale: number analyzed (Participants) | 83 | 83
  8-week: Self-Regulatory Subscale | 86.3 (17.7) | 82.5 (21.6)
  6-month: Self-Regulatory Subscale: number analyzed (Participants) | 83 | 79
  6-month: Self-Regulatory Subscale | 84.4 (23.0) | 83.1 (20.4)
  Baseline: Exercise Subscale | 84.8 (16.8) | 83.9 (18.5)
  8-week: Exercise Subscale: number analyzed (Participants) | 83 | 83
  8-week: Exercise Subscale | 87.8 (14.3) | 84.9 (20.5)
  6-month Exercise Subscale: number analyzed (Participants) | 83 | 79
  6-month Exercise Subscale | 80.3 (21.8) | 77.7 (24.2)

12. Secondary Outcome: Hip Disability and Osteoarthritis Outcome Score (HOOS)
Description: A 40-item questionnaire that contains five domains (symptoms, pain, activity of daily living (ADL), sport and recreation, and quality of life). Each scale ranges from 0-100, where higher scores are better, indicating lower hip-related disability.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
score on a scale
  Baseline Symptoms | 67.8 (18.3) | 68.6 (15.0)
  8-weeks Symptoms: number analyzed (Participants) | 83 | 83
  8-weeks Symptoms | 80.6 (12.8) | 77.4 (15.6)
  6-months Symptoms: number analyzed (Participants) | 83 | 79
  6-months Symptoms | 80.4 (13.6) | 81.6 (15.5)
  Baseline Pain | 56.1 (12.4) | 57.7 (11.4)
  8-weeks Pain: number analyzed (Participants) | 83 | 83
  8-weeks Pain | 73.8 (13.7) | 71.9 (17.2)
  6-months Pain: number analyzed (Participants) | 83 | 79
  6-months Pain | 74.1 (15.6) | 76.5 (17.1)
  Baseline ADL | 64.9 (16.7) | 66.0 (16.6)
  8-weeks ADL: number analyzed (Participants) | 83 | 83
  8-weeks ADL | 81.1 (13.9) | 78.1 (16.2)
  6-months ADL: number analyzed (Participants) | 83 | 79
  6-months ADL | 80.3 (15.1) | 80.6 (16.9)
  Baseline Sports | 50.3 (23.7) | 48.5 (24.7)
  8-weeks Sports: number analyzed (Participants) | 83 | 83
  8-weeks Sports | 70.7 (19.9) | 64.2 (24.7)
  6-months Sports: number analyzed (Participants) | 83 | 79
  6-months Sports | 68.6 (23.6) | 66.2 (27.4)
  Baseline Quality of life | 48.9 (19.8) | 51.9 (18.3)
  8-weeks Quality of Life: number analyzed (Participants) | 83 | 83
  8-weeks Quality of Life | 63.9 (18.6) | 62.6 (21.4)
  6-months Quality of Life: number analyzed (Participants) | 83 | 79
  6-months Quality of Life | 64.9 (20.6) | 70.0 (21.2)

13. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS)-29
Description: A 29-item short form questionnaire developed by the National Institutes of Health that assesses the following domains of health-related quality of life: physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, and pain intensity. Higher scores indicate better greater presence of each outcome. Possible T-scores for each domain as follows, where a T-score of 50 equals the mean of the United States population and every 10 points above or below the mean is 1 standard deviation away (e.g., a 60 is 1 standard deviation above the mean):
  Physical Function: 22.5-57.0; Anxiety: 40.3-81.6; Depression: 41.0-79.4; Fatigue: 33.7-75.8; Sleep Disturbance: 32.0-73.3; Social Roles: 27.5-64.2; Pain Interference: 41.6-75.6.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
T-Score
  Physical function--Baseline | 41.8 (5.6) | 42.1 (6.1)
  Physical function--8-weeks: number analyzed (Participants) | 83 | 83
  Physical function--8-weeks | 46.2 (6.4) | 44.5 (7.3)
  Physical function--6-months: number analyzed (Participants) | 83 | 79
  Physical function--6-months | 46.5 (7.2) | 45.3 (7.0)
  Anxiety--Baseline | 48.4 (8.4) | 46.0 (8.1)
  Anxiety--8-weeks: number analyzed (Participants) | 83 | 83
  Anxiety--8-weeks | 45.0 (6.9) | 45.8 (8.1)
  Anxiety--6-months: number analyzed (Participants) | 83 | 79
  Anxiety--6-months | 45.4 (7.2) | 44.1 (6.7)
  Depression--Baseline | 46.3 (6.8) | 45.3 (6.8)
  Depression--8-weeks: number analyzed (Participants) | 83 | 83
  Depression--8-weeks | 43.9 (5.9) | 45.6 (7.5)
  Depression--6-months: number analyzed (Participants) | 83 | 79
  Depression--6-months | 44.3 (5.9) | 44.8 (6.7)
  Fatigue--Baseline | 47.4 (7.9) | 47.6 (8.8)
  Fatigue--8-weeks: number analyzed (Participants) | 83 | 83
  Fatigue--8-weeks | 45.5 (8.2) | 46.4 (8.3)
  Fatigue--6-months: number analyzed (Participants) | 83 | 79
  Fatigue--6-months | 44.5 (8.8) | 45.7 (9.3)
  Sleep Disturbance--Baseline | 51.2 (8.2) | 49.2 (7.9)
  Sleep Disturbance--8-weeks: number analyzed (Participants) | 83 | 83
  Sleep Disturbance--8-weeks | 47.3 (7.9) | 48.7 (7.4)
  Sleep Disturbance--6-months: number analyzed (Participants) | 83 | 79
  Sleep Disturbance--6-months | 48.4 (8.2) | 47.9 (8.5)
  Social Roles--Baseline | 50.3 (7.7) | 51.5 (8.6)
  Social Roles--8-weeks: number analyzed (Participants) | 83 | 83
  Social Roles--8-weeks | 53.9 (7.6) | 52.8 (7.9)
  Social Roles--6-months: number analyzed (Participants) | 83 | 79
  Social Roles--6-months | 53.8 (8.7) | 54.3 (8.5)
  Pain Interference--Baseline | 58.8 (4.8) | 58.3 (5.4)
  Pain Interference--8-weeks: number analyzed (Participants) | 83 | 83
  Pain Interference--8-weeks | 53.9 (6.5) | 55.7 (6.7)
  Pain Interference--6-months: number analyzed (Participants) | 83 | 79
  Pain Interference--6-months | 54.3 (7.5) | 53.4 (8.2)

14. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: A 13-item questionnaire that that assesses how a person perceives pain. Items can be scored as three subscales to evaluate constructs of rumination, magnification, and helplessness. Higher scores (scale of 0-52) indicate greater levels of pain catastrophizing.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
score on a scale
  Baseline | 11.8 (9.4) | 9.5 (9.2)
  8 weeks (post-intervention): number analyzed (Participants) | 83 | 83
  8 weeks (post-intervention) | 7.1 (6.7) | 6.6 (7.9)
  6-months (final assessment): number analyzed (Participants) | 83 | 79
  6-months (final assessment) | 5.5 (6.6) | 5.9 (8.0)

15. Secondary Outcome: Hip Strength
Description: A series of strength testing measurements will be conducted using a hand-held dynamometer. All participant and examiner body positions are standardized using study protocols, and measurement locations are standardized using anatomical landmarks. Strength measurements (in kilograms) are taken for the following hip motions: abduction, extension, external rotation, internal rotation, and flexion. Measurements from the weaker side were normalized to, i.e., divided by, body weight (in kilograms), therefore, there is no unit for the measure.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: unitless (kg/kg)
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
unitless (kg/kg)
  Hip Internal rotation--Baseline | 0.071 (0.027) | 0.069 (0.028)
  Hip Internal rotation--8-weeks: number analyzed (Participants) | 78 | 77
  Hip Internal rotation--8-weeks | 0.077 (0.029) | 0.069 (0.030)
  Hip Internal rotation--6-months: number analyzed (Participants) | 67 | 69
  Hip Internal rotation--6-months | 0.078 (0.029) | 0.074 (0.041)
  Hip External rotation--baseline: number analyzed (Participants) | 91 | 92
  Hip External rotation--baseline | 0.09 (0.033) | 0.089 (0.033)
  Hip External rotation--8-weeks: number analyzed (Participants) | 78 | 77
  Hip External rotation--8-weeks | 0.11 (0.037) | 0.095 (0.033)
  Hip External rotation--6-months: number analyzed (Participants) | 67 | 69
  Hip External rotation--6-months | 0.11 (0.035) | 0.092 (0.031)
  Hip Extension--baseline | 0.12 (0.060) | 0.10 (0.055)
  Hip Extension--8-weeks: number analyzed (Participants) | 78 | 77
  Hip Extension--8-weeks | 0.14 (0.067) | 0.12 (0.058)
  Hip Extension--6-months: number analyzed (Participants) | 67 | 68
  Hip Extension--6-months | 0.15 (0.067) | 0.12 (0.060)
  Hip Abduction--Baseline | 0.084 (0.033) | 0.079 (0.031)
  Hip Abduction--8-weeks: number analyzed (Participants) | 78 | 77
  Hip Abduction--8-weeks | 0.093 (0.031) | 0.086 (0.032)
  Hip Abduction--6-months: number analyzed (Participants) | 67 | 68
  Hip Abduction--6-months | 0.100 (0.035) | 0.088 (0.032)
  Hip Flexion--Baseline: number analyzed (Participants) | 91 | 92
  Hip Flexion--Baseline | 0.159 (0.063) | 0.158 (0.067)
  Hip Flexion--8-weeks: number analyzed (Participants) | 78 | 77
  Hip Flexion--8-weeks | 0.177 (0.061) | 0.172 (0.066)
  Hip Flexion--6-months: number analyzed (Participants) | 67 | 70
  Hip Flexion--6-months | 0.192 (0.065) | 0.172 (0.061)

16. Secondary Outcome: Quantitative Sensory Testing
Description: A test where the assessor uses an algometer (i.e., handheld device that calculates the amount of force applied to the skin) to measure pressure pain sensitivity at 4 sites: upper trapezius, posterior superior iliac spine, greater trochanter, and tibialis anterior; higher values indicate higher pain thresholds, with values ranging from 0 to 10.1, where 10.1 indicates the participant tolerated 10 kilograms of force/cm squared without pain and therefore, no further pressure was applied. Pressure starts at 0.00 kilograms-of-force per square centimeter and is increased by 1-kgf/cm squared per second until the participant first experiences pain.
Time Frame: Baseline, 8-weeks (i.e. post-intervention), and 6-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kgf/cm squared
Arm/Group | Hip-focused | Spine-focused
Number analyzed (Participants) | 91 | 93
kgf/cm squared
  Right Upper trapezius--baseline | 4.27 (2.17) | 4.46 (2.25)
  Right Upper trapezius--8-weeks: number analyzed (Participants) | 78 | 77
  Right Upper trapezius--8-weeks | 4.59 (1.95) | 4.50 (2.14)
  Right Upper trapezius--6-months: number analyzed (Participants) | 67 | 70
  Right Upper trapezius--6-months | 4.22 (1.84) | 4.45 (2.15)
  Right Posterior Superior Iliac Spine--baseline | 4.76 (2.29) | 5.08 (2.51)
  Right Posterior Superior Iliac Spine--8-weeks: number analyzed (Participants) | 78 | 77
  Right Posterior Superior Iliac Spine--8-weeks | 5.34 (2.25) | 5.79 (2.34)
  Right Posterior Superior Iliac Spine--6-months: number analyzed (Participants) | 67 | 70
  Right Posterior Superior Iliac Spine--6-months | 5.43 (2.33) | 5.33 (2.42)
  Right Greater trochanter--baseline | 5.48 (2.61) | 5.87 (2.79)
  Right Greater trochanter--8-weeks: number analyzed (Participants) | 78 | 77
  Right Greater trochanter--8-weeks | 6.03 (2.33) | 6.20 (2.61)
  Right Greater trochanter--6-months: number analyzed (Participants) | 67 | 70
  Right Greater trochanter--6-months | 6.05 (2.65) | 6.11 (2.54)
  Right Anterior tibialis--baseline | 4.79 (2.47) | 4.81 (2.45)
  Right Anterior tibialis--8-weeks: number analyzed (Participants) | 78 | 77
  Right Anterior tibialis--8-weeks | 5.32 (2.39) | 5.07 (2.57)
  Right Anterior tibialis--6-months: number analyzed (Participants) | 67 | 70
  Right Anterior tibialis--6-months | 5.12 (2.58) | 4.85 (2.40)
  Left Upper trapezius--baseline | 4.09 (2.24) | 4.40 (2.44)
  Left Upper trapezius--8-weeks: number analyzed (Participants) | 78 | 77
  Left Upper trapezius--8-weeks | 4.39 (1.93) | 4.37 (2.06)
  Left Upper trapezius--6-months: number analyzed (Participants) | 67 | 70
  Left Upper trapezius--6-months | 4.19 (1.84) | 4.40 (2.24)
  Left Posterior Superior Iliac Spine--baseline | 4.93 (2.45) | 5.03 (2.50)
  Left Posterior Superior Iliac Spine--8-weeks: number analyzed (Participants) | 78 | 77
  Left Posterior Superior Iliac Spine--8-weeks | 5.52 (2.33) | 5.59 (2.39)
  Left Posterior Superior Iliac Spine--6-months: number analyzed (Participants) | 67 | 70
  Left Posterior Superior Iliac Spine--6-months | 5.57 (2.44) | 5.43 (2.47)
  Left Greater trochanter--baseline | 5.46 (2.63) | 5.73 (2.80)
  Left Greater trochanter--8-weeks: number analyzed (Participants) | 78 | 77
  Left Greater trochanter--8-weeks | 6.35 (2.34) | 6.09 (2.58)
  Left Greater trochanter--6-months: number analyzed (Participants) | 67 | 70
  Left Greater trochanter--6-months | 6.00 (2.71) | 6.04 (2.69)
  Left Anterior tibialis--baseline | 4.77 (2.55) | 4.55 (2.46)
  Left Anterior tibialis--8-weeks: number analyzed (Participants) | 78 | 77
  Left Anterior tibialis--8-weeks | 5.31 (2.43) | 4.85 (2.51)
  Left Anterior tibialis--6-months: number analyzed (Participants) | 67 | 70
  Left Anterior tibialis--6-months | 5.07 (2.65) | 4.66 (2.38)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline to the 6-month post-baseline final assessment.
Description: Our definitions of adverse events and/or serious adverse events does not differ from the clinicaltrials.gov definitions.
Arm/Group | Hip-focused | Spine-focused
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/93
Serious Adverse Events (participants affected / at risk) | 9/91 | 4/93
Other Adverse Events (participants affected / at risk) | 47/91 | 39/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hip-focused (N=91) | Spine-focused (N=93)
Surgical and Medical Procedures-other, specify (Surgical and medical procedures) | 2 (2) | 1 (1) — Hip-focused Group: 1 participant had a pacemaker implanted and 1 participant had a hernia repair surgery. Spine-focused Group: 1 participant had outpatient elbow surgery. None were related to research participation.
Chest Pain (Cardiac disorders) | 2 (2) | 0 (0) — Adverse events were unrelated to research participation.
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1) — Adverse events were unrelated to research participation.
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Adverse event was unrelated to research participation.
Cardiac Disorders-others, specify (Cardiac disorders) | 1 (1) | 0 (0) — Stent placement unrelated to research participation. Note that this participant also reported heart failure ~2 months prior, which is why there are 10 events for 9 participants in the hip-focused group.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Adverse event unrelated to research participation.
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) — Adverse event unrelated to research participation.
Respiratory, Thoracic and Mediastinal Disorders-other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — COVID-19 hospitalization. Adverse event was unrelated to research participation.
Skin Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Adverse event was unrelated to research participation.
Tremor (Nervous system disorders) | 0 (0) | 1 (1) — Adverse event unrelated to research participation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hip-focused (N=91) | Spine-focused (N=93)
Fall (Injury, poisoning and procedural complications) | 9 (9) | 6 (7) — Hip-focused Group: 8 falls unrelated and 1 fall unlikely related to research participation. Spine-focused Group: 6 falls unrelated and 1 fall unlikely related to research participation.
Surgical and medical procedures-other, specify (Surgical and medical procedures) | 6 (7) | 6 (6) — All adverse events were classified as unrelated or unlikely related to research participation. Events included hip, shoulder, and spine injections; arterial and ophthalmological procedures; and dermatological, hand, knee, and prostate surgeries.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (26) | 17 (23) — Hip-focused Group: 4 adverse events were unrelated to research, 10 were unlikely related, 11 were possibly related, and 1 was probably related. Spine-focused: 3 adverse events were unrelated, 12 were unlikely related, and 8 were possibly related.
Back pain (Musculoskeletal and connective tissue disorders) | 17 (21) | 16 (20) — Hip-focused: 3 events were unrelated, 6 were unlikely related, 9 were possibly related, and 3 were definitely related to research. Spine-focused: 1 event was unrelated, 10 were unlikely related, 8 were possibly related, and 1 was definitely related.
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (15) | 13 (16) — Hip-focused Group: 5 events were unlikely related, 9 were possibly related, and 1 was probably related to research. Spine-focused Group: 4 were unrelated, 6 were unlikely related, 5 were possibly related, and 1 was definitely related to research.

LIMITATIONS AND CAVEATS:
There was no non-intervention control group in this trial. It was impossible to mask interventionists to treatment, or participants to treatment allocation. To mitigate the potential for bias, we performed treatment fidelity audits, ensuring that both groups were receiving similar levels of active intervention. The treatment delivery was resource intensive for both therapists and participants. Cost effectiveness was not evaluated as part of this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT04009837/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT04009837/ICF_000.pdf